CLINICAL TRIAL: NCT07157436
Title: Implementation of Point Of Care UltraSound in the Assessment of Crohn's Disease
Brief Title: Implementation of Point Of Care UltraSound in the Assessment of Crohn's Disease -The POCUS Study
Acronym: POCUS
Status: Terminated | Type: Observational
Why Stopped: Lack of Recruitment due to COVID-19 Pandemic (no face to face patient appointments)
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 21GA005
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2021-06

CONDITIONS: Crohn Disease of Small Intestine
Keywords: Ultrasound; Service Improvement
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Qualitative interview study: • One of the following roles:
  * NHS Gastroenterology consultant
  * NHS IBD Nurse Specialist
  * NHS Consultant Radiologist
  * NHS business managers working in gastrointestinal services
  * Patient under the care of the NHS for small bowel CD.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — observational study. non-interventional

SUMMARY:
1. Explore Stakeholder perceptions of POCUS service development and implementation in the NHS in an interview Sub-study. We will assess whether stakeholders:

   * Recognise the potential of POCUS for the management of small bowel CD;
   * feel that it should be integrated into local services;
   * feel that they have the skills/resources to deliver POCUS;
   * can establish criteria for the service success of POCUS.
2. Compare the impact of POCUS and MRE on the nature of decision-making of consultant gastroenterologists and their confidence in clinical decision making.
3. Undertake care pathway analyses of POCUS and MRE service for IBD outpatients with small bowel CD.

DETAILED DESCRIPTION:
To demonstrate feasibility of implementing POCUS for the diagnosis and management of small bowel CD in adult ambulatory IBD care and identify the barriers for wide-spread NHS adoption

Objectives:

1. Explore Stakeholder perceptions of anticipated barriers and enablers to POCUS service development and implementation
2. Compare the impact of POCUS and MRE on the nature of decision-making of consultant gastroenterologists and their confidence in clinical decision making.
3. Undertake care pathway analyses of POCUS and MRE service for IBD outpatients with small bowel CD.

Outcome:

To create an implementation toolkit to facilitate widespread POCUS adoption and integration within NHS IBD clinical practice.

1. Qualitative interview study:

   Inclusion criteria
   * Able to give valid informed consent
   * Aged 18 years or over.
   * One of the following roles

     * NHS Gastroenterology consultant
     * NHS IBD Nurse Specialist
     * NHS Consultant Radiologist
     * NHS business managers working in gastrointestinal services
     * Patient under the care of the NHS for small bowel CD. Exclusion criteria
   * Unable to communicate clearly in verbal and written English.
2. Clinical Decision-making study Inclusion criteria

   * Ability to give informed consent.
   * Full time NHS Consultant Gastroenterologist (on GMC specialist register).
   * Agreement to comply with the study training requirements, protocol and regulatory/ sponsor stipulations.
   * Have access to local Point Of Care UltraSound (POCUS) and Magnetic Resonance Enterography (MRE) services Exclusion criteria
   * Unable to access REDCap* eCRF via NHS servers. * https://projectredcap.org/software/

ELIGIBILITY:
1. Qualitative interview study:

   Inclusion criteria
   * Able to give valid informed consent
   * Aged 18 years or over.
   * One of the following roles

     * NHS Gastroenterology consultant
     * NHS IBD Nurse Specialist
     * NHS Consultant Radiologist
     * NHS business managers working in gastrointestinal services
     * Patient under the care of the NHS for small bowel CD. Exclusion criteria
   * Unable to communicate clearly in verbal and written English.
2. Clinical Decision-making study Inclusion criteria

   * Ability to give informed consent.
   * Full time NHS Consultant Gastroenterologist (on GMC specialist register).
   * Agreement to comply with the study training requirements, protocol and regulatory/ sponsor stipulations.
   * Have access to local Point Of Care UltraSound (POCUS) and Magnetic Resonance Enterography (MRE) services Exclusion criteria
   * Unable to access REDCap* eCRF via NHS servers. * https://projectredcap.org/software/

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One of the following roles
  * NHS Gastroenterology consultant
  * NHS IBD Nurse Specialist
  * NHS Consultant Radiologist
  * NHS business managers working in gastrointestinal services
  * Patient under the care of the NHS for small bowel CD.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
To create an implementation toolkit to facilitate widespread POCUS adoption and integration within NHS IBD clinical practice. | 36 months
  Total project outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham NIHR Biomedical Research Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No